CLINICAL TRIAL: NCT02230631
Title: A Survey on Hypoglycaemia Among Insulin-treated Patients With Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-4142; U1111-1147-4179 (Other: WHO)
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Part 1 (retrospective cross-sectional evaluation)
  Interventions: Other: No treatment given
- Part 2 (prospective observational evaluation)
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Two different questionnaires will be applied to patients during a regular clinical visit.

SUMMARY:
This survey is conducted in South America. The aim of this survey is to investigate hypoglycaemia among Insulin-treated patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities
* The following patients will be considered eligible for inclusion in the study: Patients with T1DM (Type 1 Diabetes Mellitus) or T2DM (Type 2 Diabetes Mellitus) treated with insulin for more than 12 months and patients at least 18 years of age at the time of the survey

Exclusion Criteria:

* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Illiterate patients and patients otherwise unable to complete a written survey
* Non-ambulatory patients
* Simultaneous participation in any other clinical study with an investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-five sites will be selected, distributed in different regions of the country, in order to be representative of the Brazilian population.
Sampling Method: Non-Probability Sample
Enrollment: 704 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The percentage of patients experiencing at least 1 hypoglycaemic event | During 4 weeks from baseline visit

SECONDARY OUTCOMES:
Hypoglycaemic events requiring hospital admission | In the 6 months prior to (Part 1 SAQ, Self-Assessment questionnaire) and 4 weeks following (Part 2 SAQ) the baseline visit
Severe hypoglycaemic events | In the 6 months prior to (Part 1 SAQ) and 4 weeks following (Part 2 SAQ) the baseline visit
Non-severe hypoglycaemic events | In the 4 weeks prior to (Part 1 SAQ) and 4 weeks following (Part 2 SAQ) the baseline visit
Nocturnal hypoglycaemic events | In the 4 weeks prior to (Part 1 SAQ) and following (Part 2 SAQ) the baseline visit
Documented symptomatic hypoglycaemic events | In the 4 weeks following the baseline visit (Patient Diary)
Hypoglycaemic events associated with a blood glucose measurement below 56 mg/dL irrespective of symptoms | In the 4 weeks following the baseline visit (Patient Diary)
All hypoglycaemic events (any type) | In the 4 weeks prior to (Part 1 SAQ) and 4 weeks following (Part 2 SAQ) the baseline visit
Difference in the reported incidence rates of hypoglycaemia | In the 4 weeks prior to (Part 1 SAQ) versus 4 weeks following (Part 2 SAQ) the baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Säo Paulo, Brazil

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com